CLINICAL TRIAL: NCT00922649
Title: Pilot Study Assessing Insulin Pump Therapy in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Animas Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: ANM002
Record Dates: First submitted 2008-03-13; First posted 2009-06-17 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Other): Insulin pump naïve subjects with type 2 diabetes who are not achieving glycemic targets (screening A1C ≥ 7.0%) on an established regimen of ≥ 2 OAs
  Interventions: Device: Insulin Pump therapy
- B (Other): Insulin pump naïve subjects with type 2 diabetes who are not achieving glycemic targets (screening A1C ≥ 7.0%) on an established regimen of basal insulin ± OAs
  Interventions: Device: Insulin Pump therapy
- C (Other): Insulin pump naïve subjects with type 2 diabetes who are not achieving glycemic targets (screening A1C ≥ 7.0%) on an established regimen basal-bolus insulin ± OAs
  Interventions: Device: Insulin Pump therapy

INTERVENTIONS:
Device: Insulin Pump therapy — Initiation of Insulin pump therapy in patients on >2 OAs (Cohort A), basal insulin ± OAs (Cohort B), or basal-bolus insulin ± OAs (Cohort C.

SUMMARY:
16-week, open-label, multi-center pilot study. Insulin pump naïve subjects with type 2 diabetes who are not achieving glycemic targets (screening A1C ≥ 7.0%) on an established regimen of either: 1) ≥ 2 OAs (Cohort A), 2) basal insulin ± OAs (Cohort B), or 3) basal-bolus insulin ± OAs (Cohort C) will initiate basal-bolus therapy with an insulin pump using a rapid-acting insulin analog.

ELIGIBILITY:
Inclusion Criteria:

1. Is 18 to 75 years of age, inclusive;
2. Has a clinical diagnosis of type 2 diabetes mellitus;
3. Is anti-glutamic acid decarboxylase (GAD) antibody negative;
4. Has an A1C ≥ 7.0% and ≤ 10.5%;
5. Has a body mass index (BMI) ≥ 25 kg/m2 and ≤ 40 kg/m2;
6. Is treated with either ≥ 2 oral antidiabetic agents (OA) or basal insulin ± OA(s) or basal-bolus insulin ± OA(s) for at least 3 months (Subjects may also be treated with exenatide [Byetta] or pramlintide [Symlin].
7. If on concomitant metformin, has serum creatinine < 1.5 mg/dL (male) or <1.4 mg/dL (female);
8. If female, has a negative urine pregnancy test

Exclusion Criteria:

1. Has experienced recurrent severe hypoglycemia (> 2 episodes) requiring assistance during the past 6 months;
2. Has clinical cardiovascular disease (CVD) as evidenced by prior myocardial infarction, stroke, arterial revascularization and/or angina with ischemic changes on ECG at rest, changes on graded exercise test, or positive cardiac imaging test results;
3. Has abnormalities on the screening (Visit 1) 12-lead ECG that are deemed by the investigator to be clinically significant;
4. Is currently being treated with or expected to require or undergo treatment with systemic steroids by oral, intravenous, or intramuscular route or potent inhaled,intrapulmonary, intranasal, or topical steroids that are known to have a high rate of systemic absorption;
5. Currently abuses drugs or alcohol or has a history of abuse that in the investigator's opinion would cause the individual to be non-compliant;
6. Has any significant medical condition, laboratory findings, or medical history that in the investigator's opinion may affect successful completion of the study and/or personal well-being;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-02-01 (Actual); Primary Completion 2008-12-01 (Actual); Study Completion 2009-01-01 (Actual)

PRIMARY OUTCOMES:
Insulin doses at Week 16 | Week 16
  To evaluate insulin doses after 16 weeks of insulin pump therapy aimed at achieving normal or near-normal glycemic control in subjects with type 2 diabetes.This included the total daily insulin dose, basal and bolus insulin doses.
Ratio of Basal-to-Bolus Insulin Dose at Week 16 | 16 weeks
  Evaluate insulin dosing patterns after 16 weeks of insulin pump therapy aimed at safely achieving normal or near-normal glycemic control in patients with type 2 diabetes
Number of daily basal rates at Week 16 | Week 16
  To evaluate insulin dosing patterns, i.e., number of daily basal rates, after 16 weeks of insulin pump therapy aimed at achieving normal or near-normal glycemic control in subjects with type 2 diabetes.

SECONDARY OUTCOMES:
A1C (Hemoglobin A1c) | Week 16
  To evaluate the effect of 16 weeks of insulin pump therapy in subjects with type 2 diabetes on glycemic outcome
7 point profile | Week 16
  Self-monitored 7-point profiles were compared at baseline and Week 16 for each cohort and all cohorts combined.
CGM Glucose Ranges - Percent of Measurements | End of study
  The percent of glucose values within the target range of 70-180 mg/dL, as measured by CGM
Body Weight | Week 16
  Weight change was evaluated at Week 16 for each cohort and all cohorts combined.
Hypoglycemia | Week 16
  The incidence (percent of patients with at least one episode of hypoglycemia) of minor hypoglycemia was evaluated respectively. Minor hypoglycemia was defined as symptoms consistent with hypoglycemia that either resolved spontaneously or upon self-treatment with oral carbohydrate. Severe hypoglycemia referred to symptoms consistent with hypoglycemia during which the patient required the assistance of another individual and was associated with a documented glucose concentration less than 56 mg/dL or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon.
Change from baseline to week 16 in Patient Reported Outcomes (PROs) | Week 16
  PROs were assessed at Baseline, Wk 8 (except for EQ-5D) and Wk 16, including EuroQol-5 Dimensions (EQ-5D) (Generic health-related QoL), Diabetes Symptom Checklist-Revised (DSC-R) (Diabetes-specific QoL), and Insulin Delivery System Rating Questionnaire (IDSRQ) (Treatment Satisfaction with insulin delivery system)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute, Inc.; Bruce Bode, MD, Principal Investigator — Atlanta Diabetes Associates, Inc.; Mark Kipnes, MD, Principal Investigator — dgd Research, Inc.; John Liljenquist, MD, Principal Investigator — Rocky Mountain Diabetes and Osteoporosis Center, PA; Lyle Myers, M.D, Principal Investigator — Kentucky Diabetes Endocrinology Center; Sunder Mudaliar, MD, Principal Investigator — University of California, San Diego
Locations (6):
- United States (6):
  - The Regents of the University of California on behalf of its San Diego campus, La Jolla, California
  - AMCR Institute, Inc., San Diego, California
  - Atlanta Diabetes Associates, Inc., Atlanta, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, PA, Idaho Falls, Idaho
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - dgd Research, Inc., San Antonio, Texas

REFERENCES:
- [Derived] Peyrot M, Rubin RR, Chen X, Frias JP. Associations between improved glucose control and patient-reported outcomes after initiation of insulin pump therapy in patients with type 2 diabetes mellitus. Diabetes Technol Ther. 2011 Apr;13(4):471-6. doi: 10.1089/dia.2010.0167. Epub 2011 Feb 28. PMID 21355725
- [Derived] Rubin RR, Peyrot M, Chen X, Frias JP. Patient-reported outcomes from a 16-week open-label, multicenter study of insulin pump therapy in patients with type 2 diabetes mellitus. Diabetes Technol Ther. 2010 Nov;12(11):901-6. doi: 10.1089/dia.2010.0075. Epub 2010 Sep 30. PMID 20879963